CLINICAL TRIAL: NCT03138499
Title: Randomized, Open-label, Phase 3 Trial of Nivolumab Plus Brentuximab Vedotin Versus Brentuximab Vedotin Alone in Participants With Relapsed Refractory or Ineligible for Autologous Stem Cell Transplant (ASCT) Advanced Stage Classical Hodgkin Lymphoma (CheckMate 812: CHECKpoint Pathway and nivoluMAb Clinical Trial Evaluation 812)
Brief Title: A Study of Nivolumab Plus Brentuximab Vedotin Versus Brentuximab Vedotin Alone in Patients With Advanced Stage Classical Hodgkin Lymphoma, Who Are Relapsed/ Refractory or Who Are Not Eligible for Autologous Stem Cell Transplant,
Acronym: CheckMate 812
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient enrollment.
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Seagen Inc. (Industry); Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-812; 2017-000847-41 (EudraCT Number)
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Results first posted 2022-04-12 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Hodgkin's Disease
MeSH Terms: conditions — Hodgkin Disease | interventions — Nivolumab; Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Module A (Experimental): Nivolumab combined with Brentuximab
  Interventions: Biological: Nivolumab; Biological: Brentuximab vedotin
- Module B (Experimental): Brentuximab alone
  Interventions: Biological: Brentuximab vedotin

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo
  Arms: Module A
Biological: Brentuximab vedotin — Specified dose on specified days
  Other Names: Adcetris

SUMMARY:
The purpose of this study is to determine whether an investigational immuno-therapy combination, nivolumab with Brentuximab vedotin compared to Brentuximab vedotin alone is safe and effective in the treatment of relapsed and refractory Classical Hodgkin Lymphoma. The participants of this trial will comprise of patients who have relapsed or did not respond to treatment and are not eligible for stem cell transplant

ELIGIBILITY:
Inclusion Criteria

* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
* Participants must have a pathologic diagnosis of classical Hodgkin lymphoma (cHL) who are relapsed or refractory with one of the following:.

  i) Autologous stem cell transplant (ASCT) ineligible patients.

ii) Patients after failure of ASCT.

- Must have at least one lesion that is > 15 mm (1.5 cm) in the longest diameter and avid by Fluoro Deoxy Glucose (FDG) Positron Emission Tomography (PET) scan.

Exclusion Criteria

* Known central nervous system lymphoma.
* Participants with nodular lymphocyte-predominant Hodgkin lymphoma (HL).
* Participants with known history of pancreatitis or progressive multifocal leukoencephalopathy (PML).
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (22):
- United States (20):
  - City of Hope National Medical Center, Duarte, California
  - Pacific Shores Medical Group, Long Beach, California
  - University of Southern California, Los Angeles, California
  - UCLA Clinical and Translational Research Center (CTRC), Los Angeles, California
  - Local Institution, Palo Alto, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - Hartford Healthcare Cancer Institute at the Hospital of Central Connecticut, Plainville, Connecticut
  - Orlando Health, Inc, Orlando, Florida
  - Parkview Cancer Center, Fort Wayne, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Dana Farber/Harvard Cancer Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Bon Secours Saint Francis Cancer Center, Greenville, South Carolina
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center-merge, Houston, Texas
- Local Institution, Sendai, Miyagi, Japan
- Local Institution, San Juan, Puerto Rico

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 23 participants were randomized for study participation, 22 received at least 1 dose of study drug.
Groups:
- Nivolumab + Brentuximab Vedotin (BV): Nivolumab 360 mg IV every 3 weeks until progression or unacceptable toxicity (except for patients in CR who can discontinue at 2 years) plus BV 1.8 mg/kg IV every 3 weeks for up to 16 cycles, or until progression or unacceptable toxicity, whichever occurs first.
- Brentuximab Vedotin (BV): BV alone 1.8 mg/kg every 3 weeks for up to 16 cycles, or until disease progression or unacceptable toxicity, whichever occurs first
Period: Overall Study
Arm/Group | Nivolumab + Brentuximab Vedotin (BV) | Brentuximab Vedotin (BV)
Started | 12 | 11
Completed | 3 | 1
Not Completed | 9 | 10
Not completed — Lost to Follow-up | 1 | 0
Not completed — Participants withdrew consent | 1 | 0
Not completed — Participant discontinued study before treatment | 0 | 1
Not completed — Disease Progression | 2 | 6
Not completed — Study drug toxicity | 2 | 2
Not completed — Participant request to discontinue study treatment | 1 | 1
Not completed — Other reasons | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab + Brentuximab Vedotin (BV) | Brentuximab Vedotin (BV) | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.5 (13.1) | 42.3 (16.1) | 39.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 9 | 7 | 16
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE | 7 | 4 | 11
  BLACK OR AFRICAN AMERICAN | 3 | 2 | 5
  JAPANESE | 0 | 1 | 1
  ASIAN OTHER | 0 | 1 | 1
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 1 | 0 | 1
  OTHER | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS) is defined as time from date of randomization to death, or disease progression per investigator assessment estimated using the Kaplan-Meier (KM) product-limit method.
Time Frame: From randomization to date of death, or disease progression (up to approximately 45 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Brentuximab Vedotin (BV) | Brentuximab Vedotin (BV)
Number analyzed (Participants) | 12 | 11
Months | 14.32 [10.12 to NA] — Insufficient number of participants with events | 7.93 [2.86 to NA] — Insufficient number of participants with events

2. Secondary Outcome: Complete Response Rate (CRR):
Description: Complete Response Rate (CRR) is defined as the number of participants who have achieved complete response (Lugano 2014 classification) per investigator assessment. Complete response is considered a score of 1, 2, or 3.
  Per the Lugano criteria:
  Positron emission tomography (PET) negative scans are defined on the 5-point scale as scores of 1, 2, or 3 (where 1 = no uptake above background; 2 = uptake </= mediastinum; and 3 = uptake > mediastinum but </= liver) and PET-positive scans, as scores of 4 or 5 (where 4 = uptake moderately higher than liver; 5 = uptake markedly higher than liver and/or new lesions). Response on PET scans should be reported as complete metabolic response (CMR) partial metabolic response (PMR), SMD (stable metabolic disease), or PMD (progressive metabolic disease).
Time Frame: From randomization up to approximately 45 months
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Groups:
- Brentuximab Vedotin (BV): BV alone 1.8 mg/kg every 3 weeks for 16 cycles, or until progression or unacceptable toxicity, whichever occurs first
Arm/Group | Nivolumab + Brentuximab Vedotin (BV) | Brentuximab Vedotin (BV)
Number analyzed (Participants) | 12 | 11
Participants | 4 | 3

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) is defined as the number of participants with a Best Overall Response (BOR) of complete response (CR) or partial response (PR) (Lugano 2014 classification) per investigator assessment. Complete response is considered a score of 1, 2, or 3. Partial response is considered a score of 4 or 5.
  Per the Lugano criteria:
  Positron emission tomography (PET) negative scans are defined on the 5-point scale as scores of 1, 2, or 3 (where 1 = no uptake above background; 2 = uptake </= mediastinum; and 3 = uptake > mediastinum but </= liver) and PET-positive scans, as scores of 4 or 5 (where 4 = uptake moderately higher than liver; 5 = uptake markedly higher than liver and/or new lesions). Response on PET scans should be reported as complete metabolic response (CMR) partial metabolic response (PMR), SMD (stable metabolic disease), or PMD (progressive metabolic disease).
Time Frame: From randomization up to approximately 45 months
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Brentuximab Vedotin (BV) | Brentuximab Vedotin (BV)
Number analyzed (Participants) | 12 | 11
Participants | 8 | 5

4. Secondary Outcome: Duration of Response (DOR)
Description: The time from first response (Complete response (CR) or partial response (PR)) to the date of initial objectively documented progression (2014 Lugano classification) or death due to any cause per investigator assessment estimated using the Kaplan-Meier (KM) product-limit method. Complete response is considered a score of 1, 2, or 3. Partial response is considered a score of 4 or 5.
  Per the Lugano criteria:
  Positron emission tomography (PET) negative scans are defined on the 5-point scale as scores of 1, 2, or 3 (where 1 = no uptake above background; 2 = uptake </= mediastinum; and 3 = uptake > mediastinum but </= liver) and PET-positive scans, as scores of 4 or 5 (where 4 = uptake moderately higher than liver; 5 = uptake markedly higher than liver and/or new lesions). Response on PET scans should be reported as complete metabolic response (CMR) partial metabolic response (PMR), SMD (stable metabolic disease), or PMD (progressive metabolic disease).
Time Frame: From randomization to date of documented progression or death (up to approximately 45 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Brentuximab Vedotin (BV) | Brentuximab Vedotin (BV)
Number analyzed (Participants) | 8 | 5
Months | 11.27 [7.39 to 11.27] | 7.00 [1.54 to NA] — Insufficient number of participants with events

5. Secondary Outcome: Duration of Complete Response (DOCR)
Description: Duration of complete response (DOR) is defined as the time from first complete response to the date of initial objectively documented progression (2014 Lugano classification) or death due to any cause per investigator assessment estimated using the Kaplan-Meier (KM) product-limit method. Complete response is considered a score of 1, 2, or 3.
  Per the Lugano criteria:
  Positron emission tomography (PET) negative scans are defined on the 5-point scale as scores of 1, 2, or 3 (where 1 = no uptake above background; 2 = uptake </= mediastinum; and 3 = uptake > mediastinum but </= liver) and PET-positive scans, as scores of 4 or 5 (where 4 = uptake moderately higher than liver; 5 = uptake markedly higher than liver and/or new lesions). Response on PET scans should be reported as complete metabolic response (CMR) partial metabolic response (PMR), SMD (stable metabolic disease), or PMD (progressive metabolic disease).
Time Frame: From randomization to date of documented progression or death (up to approximately 45 months)
Population: All randomized participants with objective response of complete response (CR)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Brentuximab Vedotin (BV) | Brentuximab Vedotin (BV)
Number analyzed (Participants) | 4 | 3
Months | 7.85 [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

6. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time between the date of randomization and the date of death estimated using the Kaplan-Meier (KM) product-limit method
Time Frame: From randomization to the date of death (up to approximately 3 years 7 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Brentuximab Vedotin (BV) | Brentuximab Vedotin (BV)
Number analyzed (Participants) | 12 | 11
Months | NA [25.40 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: From first dose to up to 100 days post last dose (up to approximately 2 years) All-cause mortality was assessed from date of first dose to study completion (up to approximately 3 years 7 months)
Description: 23 participants were randomized for study participation, 22 received at least 1 dose of study drug and one participant discontinued study before treatment. Adverse events were collected for all treated participants who received at least 1 dose of study treatment.
Arm/Group | Nivolumab + Brentuximab Vedotin (BV) | Brentuximab Vedotin (BV)
All-Cause Mortality (participants affected / at risk) | 1/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 6/12 | 1/10
Other Adverse Events (participants affected / at risk) | 12/12 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Brentuximab Vedotin (BV) (N=12) | Brentuximab Vedotin (BV) (N=10)
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Adenovirus infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Seizure (Nervous system disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Brentuximab Vedotin (BV) (N=12) | Brentuximab Vedotin (BV) (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 2
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 3
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Eye discharge (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0
Scleral hyperaemia (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 3 | 0
Chest pain (General disorders) | 2 | 0
Chills (General disorders) | 3 | 0
Fatigue (General disorders) | 6 | 4
Influenza like illness (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 4 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 2
Abscess jaw (Infections and infestations) | 1 | 0
Body tinea (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Scrotal abscess (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Viral pericarditis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 2
Blood bilirubin decreased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 1 | 0
Breath sounds abnormal (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Influenza B virus test positive (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 2
Neutrophil count decreased (Investigations) | 2 | 2
Platelet count decreased (Investigations) | 1 | 1
Weight decreased (Investigations) | 2 | 1
Weight increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 2
Neuropathy peripheral (Nervous system disorders) | 6 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 1
Anxiety (Psychiatric disorders) | 3 | 1
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urine odour abnormal (Renal and urinary disorders) | 1 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Due to a treatment paradigm shift and subsequent low enrollment, the Sponsor chose to terminate the study and consequently there is limited data. These reasons were unrelated to any adverse events (AEs) or safety concerns.

The sample size was smaller than expected, therefore, results should be interpreted with caution. PFS, CRR, and ORR outcomes should be interpreted with caution given large confidence intervals around medians and early study closure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT03138499/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT03138499/SAP_001.pdf